CLINICAL TRIAL: NCT00850460
Title: Quality of Life and Metabolic Alterations in Patients With Statin-Associated Myopathy
Brief Title: Quality of Life in Patients With Statin-Associated Myopathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator left institution and no PI has been found to continue the study
Sponsor: Rockefeller University (Other)
Collaborators: Cornell University (Other); Adelphi University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: PAM-0655
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Statin Adverse Reaction
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Simvastatin; Pravastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Lactose placebo pill
  Interventions: Drug: Placebo
- Statins (Active Comparator): Statin medications
  Interventions: Drug: Statins

INTERVENTIONS:
Drug: Statins — Subjects will be randomized to continue their statin dosage or placebo for 8 weeks. They will stay on the same dosage as prescribed by their physician. Usual dosage for atorvastatin 10-80 mg/tab once daily by mouth; simvastatin 20-80 mg/tab once daily by mouth; pravastatin 10-80 mg/tab once daily by mouth; rosuvastatin 5-20 mg/tab once daily by mouth.
  Other Names: atorvastatin, simvastatin, pravastatin, rosuvastatin
  Arms: Statins
Drug: Placebo — Placebo pills will consist of lactose and will be given one capsule once daily
  Other Names: lactose pills
  Arms: Placebo

SUMMARY:
The proposed study will focus on possible effects of statins on muscle strength and why they become tired more easily, quality of life, and measurements to understand why muscles are not able to fully utilize fats. The investigators are specifically interested in statin users and the impact of muscle symptoms on daily activities and quality of life.

This study hypothesize that patients with likely statin-associated myopathy have a metabolic dysregulation in fuel utilization such that compared to patients continuing statins, those on placebo will show:

1. improved Individualized Neuromuscular Quality of Life (INQoL) and Short Form-36 (SF-36) scores (primary end point)
2. alleviation of muscle symptoms,
3. increased utilization of fatty acids as a fuel source reflected by the metabolic test results
4. decreased intramyocellular lipid (IMCL)
5. improved insulin sensitivity.

DETAILED DESCRIPTION:
The proposed study will focus on possible effects of statins on muscle strength and quality of life, and measurements to understand why muscles of statin users are not able to fully utilize fats. The investigators are specifically interested in statin users and the impact of muscle symptoms on daily activities and quality of life.

This study hypothesizes that patients with likely statin-associated myopathy have a metabolic dysregulation in fuel utilization such that compared to patients continuing statins, those on placebo will show:

1. improved INQoL and SF-36 scores (primary end point)
2. alleviation of muscle symptoms,
3. increased utilization of fatty acids as a fuel source reflected by the metabolic test results
4. decreased IMCL
5. improved insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* males and females 30-60 yrs old
* experiencing muscle pain, weakness, numbness or cramping that they perceive to interfere with activities of daily living (ADLs), but able to ambulate independently (in order to perform exercise tests)
* muscle symptoms started/ occurred within one year of starting statin treatment or within one year of changing statin brand or dose adjustment
* currently taking a statin (has been taking medications ≥ 80% of the time or at least 5 days/week)
* ≤ 15% probability of having a cardiovascular (CV) event in the next 10 years calculated using an online CV risk calculator (while on current statin) for the questionnaire portion; AND with a low or a moderate American College of Sports Medicine (ACSM) risk stratification for a cardiovascular event during a treadmill test for the full metabolic study
* must agree to have a letter sent to inform the health care provider who prescribed the statin of study participation except for subjects referred by Metropolitan Hospital physicians

Exclusion Criteria:

* concomitant treatment with other lipid-lowering agents
* impaired liver or kidney function ( alanine aminotransferase (ALT) or asparate aminotransferase (AST) ≥ 3x upper limit of normal, creatinine ≥ 3x or creatine phosphokinase (CPK) ≥ 5x upper limit of normal)
* untreated hypo or hyperthyroidism
* current treatment with other medications known to increase risk of myopathy (e.g. cyclosporine, azithromycin, erythromycin and other macrolide antibiotics, azole antifungals, fusidic acid, digoxin)
* documented history of muscle disorder or myopathy other than statin-associated myopathy
* anemia (Hb< 110 g/dL)
* cancer within 5 years of enrollment except basal or squamous cell carcinoma (CA) of the skin
* diabetes
* HIV-1 infection
* Uncontrolled blood pressure ≥ 160/100
* known coronary artery disease or peripheral vascular disease
* chronic illnesses such as lupus, rheumatoid arthritis, psoriasis
* any condition, that at the investigators' discretion would impact/ bias the study data
* long term oral, nasal, or inhaler steroid use > 6 months
* on Hormone Therapy except for thyroid replacement
* alcohol consumption ≥ 40 g/day (3 glasses/day wine or beers or binge drinking ≥ 4 glasses/night)
* engaged in significant amounts of sport or strenuous leisure activity (> 60 min four times per week)
* surgery in the past 6 months except for minor excision/incision procedures,
* 12-L electrocardiogram demonstrating old/new myocardial infarction/ ischemia or other findings that, at the cardiologist's discretion, may put the subject at high risk
* cognitive impairment that prevents comprehension of questionnaires
* inability to read English (questionnaire language)

Exclusions for the metabolic study:

* currently taking beta blockers
* body mass index > 28 kg/m2
* premenopausal females < 50 yrs (menopause defined as 12 consecutive months without menstruation (in order to avoid the confounding effect of the menstrual cycle phase on fuel selection)
* physical disability or previous injury that prevents safe exercise testing
* do not meet the magnetic resonance spectroscopy (MRS) prescreening criteria

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D Maningat, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Advertisements were placed (internet, radio, print) and a screening phone questionnaire was administered by study staff to determine potential inclusion. A collaboration with the Metropolitan Hospital (NY) was also established for potential referrals.
Pre-assignment Details: Subjects in whom statins are possibly causative, using the World Health Organization (WHO)-Causality Assessment form, were invited to the outpatient clinic for 2 screening visits. Subjects found to be at high risk for cardiovascular events and those unwilling to be shifted to placebo were not enrolled.
Period: Overall Study
Arm/Group | Placebo | Statins
Started | 7 | 7
Started - Week 0 | 7 | 7
Completion - Week 8 | 3 | 3
Completed | 3 | 3
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: Males and females 30-60 years old, taking a statin, experiencing muscle pain, weakness, cramping and not at high risk for a cardiovascular event
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Statins | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Individualized Neuromuscular Quality of Life (INQoL) Mean Scores From Week 0 to Week 8
Description: Scores from the self-administered INQoL questionnaire will be compared at the start of the study (Week 0) and at the end (Week 8) between the statin-treated group and the placebo group. Scores range from 0-100, with 100 being a better outcome. Measures reported are the means of Week 0 and week 8, measures of dispersion is the range of the results (3 per group).
Time Frame: Week 0 to Week 8
Population: Three patients from each group completed the questionnaire portion of the study at Week 0 and Week 8.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Statins
Number analyzed (Participants) | 3 | 3
units on a scale
  Week 0 Mean Score | 65 [43.9 to 95] | 76 [67.2 to 81.7]
  Week 8 Mean Score | 67 [53.3 to 88.3] | 50 [43.9 to 60.6]

2. Primary Outcome: Individualized Short Form-36 (SF-36) Mean Scores (Physical Component) From Week 0 to Week 8
Description: Scores from the self-administered SF-36 (Physical component) questionnaire were measured at the start (Week 0) of the study and at the end (Week 8) among patients in the placebo- and statin-treated group. Mean scores range from 0 (minimum) - 100 (maximum) with higher mean scores reflecting better outcomes. Measures reported are the means of Week 0 and week 8, measures of dispersion is the range of scores.
Time Frame: Week 0 to Week 8
Population: Three patients from each group completed the questionnaire portion of the study at Week 0 and Week 8.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Placebo | Statins
Number analyzed (Participants) | 3 | 3
units on a scale
  Week 0 Mean Score | 50 [45.7 to 58] | 53 [49.7 to 54.4]
  Week 8 Mean Score | 56 [53.8 to 58.6] | 48 [47.3 to 48.2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the subjects were enrolled in the study until study termination (eight weeks). The study ran for two years.
Arm/Group | Placebo | Statins
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes